CLINICAL TRIAL: NCT05152888
Title: The Impact of Pcsk-9 Inhibition on PET Coronary Flow Reserve in Patients at High Cardiovascular Risk (EMPOWER Study)
Brief Title: The Impact of Pcsk-9 Inhibition on PET CFR in Patients at High CV Risk
Acronym: EMPOWER
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Diana M. Lopez, MD, Cardiologist, Brigham and Women's Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2021P003360
Record Dates: First submitted 2021-11-29; First posted 2021-12-10 (Actual); Last update posted 2025-11-04 (Actual); Status verified 2025-11

CONDITIONS: Stable Coronary Disease
MeSH Terms: interventions — evolocumab

STUDY DESIGN:
Intervention Model Description: The study protocol is an open label pilot study with a parallel control group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Evolocumab (Experimental): Informed consent will be obtained from study participants willing to participate in EMPOWER. Study participants will then undergo the baseline rest/stress cardiac PET scan along with CCTA. The final PET scan and CCTA will occur at 12 months after the intervention.
  Interventions: Drug: Evolocumab
- Control (No Intervention): Informed consent will be obtained from study participants willing to participate in EMPOWER. Study participants will then undergo the baseline rest/stress cardiac PET scan along with CCTA. The final PET scan and CCTA will occur at 12 months after the baseline.

INTERVENTIONS:
Drug: Evolocumab — Evolocumab is a human monoclonal antibody that inhibits proprotein convertase subtilisin-kexin type 9 (PCSK9). Evolocumab was FDA approved in 2015 for the treatment of hyperlipidemia and subsequently approved in 2017 for the prevention of stroke and heart attack. 140mg single use SureClick autoinjector that is administered subcutaneously once every 2 weeks.
  Other Names: Repatha
  Arms: Evolocumab

SUMMARY:
The study protocol is a single-arm, open label pilot study designed to evaluate the impact of PCSK-9 inhibition on coronary blood flow in patients with stable coronary artery disease. Patients with stable coronary artery disease will be recruited from the BWH Cardiovascular Medicine clinic and/or from the BWH Nuclear Cardiology Laboratory. A target sample size of 50 participants will undergo imaging with N-13 ammonia or Rubidium-82 positron emission tomography (PET) and coronary computed tomography angiography (CCTA) before and after 12 months of PCSK-9 inhibition with Evolocumab to assess changes in myocardial blood flow, and plaque volume. To help account for physiological changes that may occur in myocardial blood flow and inflammatory biomarkers during the study period, we will also recruit a parallel control group of stable CAD patients who will undergo similar baseline and 12-month imaging and biomarker assessment. We plan to recruit 15 patients in the parallel control group.

DETAILED DESCRIPTION:
The investigators propose an open-label investigator-initiated trial to directly test whether PCSK-9 inhibition with Evolocumab in patients with stable CAD improves PET CFR and stress MBF. To further elucidate the possible mechanisms by which myocardial blood flow improves with PCSK-9 inhibition, the investigators will assess changes in inflammatory biomarkers. The findings of this translational study will provide a physiological read-out of the comprehensive effects of Evolocumab on tissue perfusion and microvascular function in a high-risk population. As such, these data would serve to provide a mechanistic explanation for why Evolocumab may reduce cardiovascular events beyond a reduction in plaque burden and composition.

The central hypothesis of this study is that PCSK-9 inhibition will quantitatively improve myocardial blood flow as measured by positron emission tomography (PET) in patients with stable coronary artery disease. The investigators postulate that the improvement in myocardial blood flow will correlate with a reduction in inflammatory biomarkers, and not simply an improvement in coronary epicardial plaque burden.

ELIGIBILITY:
Intervention Group:

Inclusion Criteria:

* Age: ≥ 50 (men) or ≥ 55 (women)
* Low-density lipoprotein cholesterol (LDL-C) ≥ 70 mg/dL
* Stable coronary artery disease (without plan to undergo revascularization before randomization) defined as one or more of the following:

  1. Abnormal nuclear perfusion imaging

     1. At least moderate ischemia involving >10% of the LV myocardium or
     2. Global coronary flow reserve (CFR) <1.8 or
     3. Stress myocardial blood flow (MBF) <1.8
  2. Abnormal coronary angiography (invasive coronary angiography or coronary computed tomography)

     1. ≥ 50% stenosis in ≥ 2 coronary vessels or
     2. Diffuse atherosclerosis in a 3-vessel distribution
  3. Elevated coronary calcium score

     1. CAC >100 + >1 ASCVD risk factor
     2. CAC >300
* If the patient is on a statin they must be on a stable dose for at least 3 months prior to enrollment.

Exclusion Criteria:

* History of myocardial infarction or stroke
* CABG < 3 months prior to screening
* Homozygous familial hypercholesterolemia
* History of cardiac transplantation
* LV ejection fraction < 40% or New York Heart Failure Association (NYHA) class III-IV for angina and/or dyspnea.
* History of infiltrative or hypertrophic cardiomyopathy
* Severe valvular disease
* Uncontrolled or recurrent ventricular tachycardia
* Fasting triglycerides > 500 mg/dL
* GFR ˂ 30 mL/min/1.73 m²
* Current use of a PCSK-9 inhibitor
* Currently pregnant or breastfeeding
* Contraindication to receive vasodilator agent
* Latex allergy

Parallel Control Group:

Patients will be invited to participate in the parallel control group if they meet study criteria, but 1) have a latex allergy and cannot use the Evolocumab autoinjector 2) LDL-C is just below the enrollment criteria (LDL 60-69), or 3) meet study criteria but prefer to not take an injectable medication at this time.

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-03-03 (Actual); Primary Completion 2027-03-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Coronary Flow Reserve | Change (from baseline) in global CFR, as measured by PET imaging at 52 weeks after initiation of Evolocumab therapy.
  Change in global coronary flow reserve (CFR) after 12 months of therapy with Evolocumab
Stress Myocardial Blood Flow (MBF) | Change (from baseline) in stress MBF, as measured by PET imaging at 52 weeks after initiation of Evolocumab therapy.
  Change in stress Myocardial Blood Flow (MBF) after 12 months of therapy with Evolocumab

SECONDARY OUTCOMES:
Total Perfusion Deficit (TPD) | Change (from baseline) in TPD, as measured by PET imaging at 52 weeks after initiation of Evolocumab therapy.
  Change in Total Perfusion Deficit (TPD) after 12 months of therapy with Evolocumab

CONTACTS AND LOCATIONS:
Overall Officials: Diana Lopez, MD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No